CLINICAL TRIAL: NCT03814538
Title: Assessment of the Incidence of Expiratory Flow Limitation in Patients Undergoing Thoracic Surgery
Brief Title: Expiratory Flow Limitation in Thoracic Surgery (EFLinTOR)
Acronym: (EFLinTOR)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Professor, University of Parma
Other Study IDs: 876/2018/OSS/AOUPR
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Thoracic Surgery; General Anesthesia
Keywords: Postoperative pulmonary complications; Incidence of EFL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and rationale of the study: During general anesthesia, the residual functional capacity (FRC) is reduced. If the FRC is lower than the minimum volume necessary to maintain the airway opening (closing capacity, CC), a pulmonary parenchyma derecruitment leads to the phenomenon of expiratory flow limitation (EFL). In recent years, new methods are being studied to assess EFL. In the study by Marangoni E, et. al., has been shown how the sudden subtraction of 3 cmH2O to the value of the tele-expiratory positive pressure (PEEP test) is sufficient to establish the presence of the EFL.

The presence of EFL measured by this method seems to correlate, in abdominal surgery, with the development of post-operative pulmonary complications. In the area of anesthesia in thoracic surgery, neither the incidence nor the relevance of the EFL are known, so a study is needed that evaluates both.

The aim of the study is to determine the incidence of expiratory flow limitation in patients undergoing thoracic surgery and ventilated in bi and monopolmonary mode.

The protective ventilation is a mechanical ventilation with a current volume (TV) of 6-8 mL / kg among to the ideal body weight (IBW), PEEP of 3-5 cmH2O and a FiO2 <80%.

The aim of this study is to evaluate the incidence of EFL in patients undergoing thoracic surgery, planned by thoracoscopy and thoracotomy in election, and to correlate this parameter with the onset of postoperative pulmonary complications. The final aim will be to verify if it is possible to identify a better approach, through the personalization of mechanical ventilation during the surgery, to reduce mortality, morbidity and hospital stay after thoracic surgery.

DETAILED DESCRIPTION:
It's a prospective and observational study, with 100 patients that undergo thoracic surgery.

The respiratory rate will be set to maintain PaCO2 at values close to eucapnia.

Controlled pressure ventilation (Pinsp ≤ 35 cmH2O) will be used only if the maximum airway pressures are reached and exceeded with controlled ventilation.

The inspiratory mixture will consist of O2: Air and possibly the halogenated anesthetic.

At the end of the operation, the patients will be transferred to Intensive Care Unit for post-operative monitoring. During the transfer will be supported with mechanical ventilation manually performed by the Anesthesiologist.

The extubation will be performed in TICCH, according to the practice of the center.

Patients will be asked to join the study by giving informed consent.

The data will be collected through a special data collection form (Case Report Form, CRF).

The following information will be collected:

In the section dedicated to the preoperative patient data will be inserted related to:

* age, weight, height, sex;
* general health conditions
* previous and concurrent diseases
* positive respiratory history for: previous pleuro-parenchymal diseases in the 30 days prior to surgery, previous interventions on the thorax, pleura or lung, presence of pleural effusion; asthma; Chronic obstructive pulmonary disease.
* history of cigarette smoking: active smoker (number of cigarettes), ex-smoker or non-smoker;
* Preoperative Therapy
* SpO2, PaO2, PaO2 / FiO2, PaCO2 (if available);
* cardiological anamnesis (echocardiography, ECG, etc.) other medical information relevant to the study

The following data will be collected on the intra-operative card:

* incidence of EFL and respiratory mechanics parameters, collected by the ventilator;
* type of surgical intervention;
* transfusion of blood derivatives;
* eventual administration of cardio / vasoactive drugs;
* duration of the surgery; other information related to the intra-operative relevant for the purpose of the study

The EFL will be registered at the following time-points:

* after the induction of anesthesia;
* after lateral positioning of the patient;
* start of One Lung Ventilation;
* 5 ' after cutting skin;
* 30 ' after cutting skin;
* 5 ' after closing skin;
* Bipulmonary ventilation;
* Positioning of the back of the patient.

The following data will be recorded in the postoperative card:

* Post-operative mechanical ventilation time
* postoperative respiratory complications;
* postoperative non-respiratory (cardiovascular, infectious, renal, surgical) complications;
* need for re-intubation in the postoperative period;
* need for ventilatory support (non-invasive ventilation, invasive ventilation) in the postoperative period;
* need for hospitalization in intensive care (expected, unexpected, cause of hospitalization, length of stay);
* duration of hospital stay; other postoperative information relevant for the purpose of the study.

Data will be analyzed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* signed informed consent
* elective thoracic surgery
* planned thoracic surgery with thoracotomy and thoracosthomy

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Patients undergoing emergency or emergency surgery
* Patients underwent cardiac and surgery
* patients underwent thoracic surgery with median sthernotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non critical ill patients (with no high risk of desaturation) undergoing general anesthesia before elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of EFL | From the induction of general anesthesia, until the end of the surgical procedure, up to 10 hours
  Evaluate the incidence of the EFL in patients undergoing thoracic surgery
Incidence of postoperative pulmonary complications (PPC) related to EFL | From immediately after surgery until hospital discharge, up to 26 weeks
  Evaluate the relationship between the incidence of EFL and the onset of PPC in patients undergoing thoracic surgery

SECONDARY OUTCOMES:
Incidence of length of in-hospital stay | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of Intensive Care Unit admission and its duration | From immediately after surgery until hospital discharge, up to 26 weeks
Duration of mechanical ventilation | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of cardiovascular postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of neurological postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of surgical postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of mortality | From immediately after surgery until hospital discharge, up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michela Tosi, MD, Principal Investigator — University of Parma; Benedetta Siroli, MD, Principal Investigator — University of Parma; Samantha Gorgoglione, MD, Principal Investigator — University of Parma; Valentina Bellini, MD, Principal Investigator — University of Parma; Anna Cozzolino, MD, Principal Investigator — University of Parma; Cristina Montanino, MD, Principal Investigator — University of Parma
Locations (1):
- Azienda Ospedaliera-Universitaria di Parma, Parma, Italy